CLINICAL TRIAL: NCT01705834
Title: The Evaluation of a Dataglove to Measure Joint Stiffness in Patients With Arthritis
Brief Title: Dataglove to Measure Joint Stiffness in Patients With Arthritis
Status: Withdrawn | Type: Observational
Why Stopped: The study protocol has been replaced with a two-glove protocol NCT02026245
Sponsor: Western Health and Social Care Trust (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Dr Philip Gardiner, Consultant Rheumatologist, Western Health and Social Care Trust
Other Study IDs: Dataglove-01
Record Dates: First submitted 2012-10-04; First posted 2012-10-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis; Stiffness; Range of movement; Goniometry; Digital; Dataglove; Outcome
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arthritis patients: Patients with Rheumatoid Arthritis

SUMMARY:
This study will investigate if an electronic dataglove can be used to measure joint stiffness in patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
We will use a dataglove to record joint movements in a small number of patients with rheumatoid arthritis. The aim of the study is to find out if changes in dynamic movements measured by the glove will correlate with symptoms of joint stiffness in the hands of patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 80
* Diagnosis of Rheumatoid arthritis
* Patients who have significant pain and stiffness in their hands
* Correct hand size to achieve a good fit to the dataglove
* Able to follow instructions for use of dataglove/computer

Exclusion Criteria:

* Severe pain in the right hand
* Severe swelling in the right hand (rated as such by the investigator)
* Severe permanent deformity or loss of function in the fingers of the right hand
* Broken or infected skin in the right hand
* Known to have been MRSA positive currently or in the past
* Unable to don and doff the disposable lining glove and the dataglove without significant discomfort
* Poor fit for the disposable lining glove or the dataglove
* History of latex allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid arthritis causing pain and stiffness in their hands.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Correlation between maximum velocity of movement and the patient reported severity of joint stiffness | Maximum of 7 days
  A significant inverse correlation is expected to be found between the patient's assessment of the severity and/or duration of stiffness and the maximum velocity of movement at the main finger joints.

SECONDARY OUTCOMES:
Number of patients withdrawing from the study | Over the period of testing of the dataglove - 7 day timeframe
  We are expecting that no more than 30% of patients will withdraw from the study due to discomfort fitting or using the dataglove.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gardiner, MB BCh BAO MD, Study Chair — Western Health and Social Services Trust; Kevin Curran, PhD, Principal Investigator — University of Ulster; Joan Condell, PhD, Principal Investigator — University of Ulster; James Connolly, BSc, Principal Investigator — University of Ulster
Locations (1):
- Department of Rheumatology, Altnagelvin Hospital, Londonderry, N.Ireland, United Kingdom